CLINICAL TRIAL: NCT04786626
Title: Ultrasound Evaluation of Uterine Healing After Vaginal Repair of Cesarean Scar Defect (CSD)
Acronym: CSD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-002
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-01

CONDITIONS: Ultrasound Evaluation
Keywords: ultrasound; cesarean scar defects; vaginal repair; resistance index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound evaluation — After vaginal, all patients were followed by traditional 2D US scanning and Doppler velocimetry on Days: 0, 2, 30, 60 and 90. Authors evaluated: scar diameter and Doppler velocimetry and resistance index (RI) of the uterine arteries, at their ascending branch

SUMMARY:
Cesarean scar defect is one of the complications after cesarean section (CSD). CSD may be further caused many long term complications, such as abnormal uterine bleeding, infertility, uterine scar pregnancy and uterine rupture. Vaginal repair due to CSDs is a minimally invasive and effective method that maintains fertility. The main concern linked to surgery is the quality of healing of the myometrial incision. However, no diagnostic method has yet been widely accepted to assess the healing process. Thus, the authors investigated uterine healing after vaginal repair with two-dimensional (2D) power Doppler ultrasound (PDU) in this study.

DETAILED DESCRIPTION:
The inclusion criteria were CSD patients who had one or more cesarean deliveries, patients who had intermenstrual spotting after the cesarean section or those in which the thickness of the residual myometrium (TRM) was less than 3.0 mm at the preoperative stage.

Patients who had a history of endocrine disorders, coagulation disorders, use of intrauterine devices, sub-mucous myoma, endometrial diseases, endometrial cysts, uterine fibroids, and adenomyosis after cesarean section were excluded from this study.

After vaginal repair, all patients were followed by traditional 2D US scanning and Doppler velocimetry on Days: 0, 2, 30, 60 and 90. Authors evaluated: scar diameter and Doppler velocimetry and resistance index (RI) of the uterine arteries, at their ascending branch.

ELIGIBILITY:
Inclusion Criteria:

1. have one or more cesarean deliveries,
2. have intermenstrual spotting after the cesarean section or TRM was less than 3.0 mm at the preoperative stage
3. underwent MRI and TVS to evaluate the size of the defect and the TRM before surgery
4. have vaginal repair of CSD
5. write consent for operation.

Exclusion Criteria:

1. have a history of endocrine disorders
2. have coagulation disorders
3. use of intrauterine devices
4. have sub-mucous myoma
5. have endometrial diseases
6. have endometrial cysts, uterine fibroids, and adenomyosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CSD patients who had one or more cesarean deliveries, patients who had intermenstrual spotting after the cesarean section or those in which the TRM was less than 3.0 mm at the preoperative stage.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-20 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Evaluation | Change from Baseline Systolic Blood Pressure at 6 months
  resistance index (RI) of the uterine arteries

SECONDARY OUTCOMES:
the size of CSD | on Days: 0, 2, 30, 60 and 90
  the length in millimeters, the width in millimeters and the depth in millimeters of CSD
the TRM of scar | on Days: 0, 2, 30, 60 and 90
  the TRM of scar

OTHER OUTCOMES:
reproductive information | 2 years
  reproductive information by questionnaire, including abortion, delivery, childbirth, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China